CLINICAL TRIAL: NCT02697812
Title: Does the Speed of Sternal Retraction During Coronary Artery Bypass Graft Surgery Affect Postoperative Pain Outcomes: A Randomized Controlled Trial
Brief Title: Does the Speed of Sternal Retraction Affect Postoperative Pain Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Tarit Saha (Other)
Responsible Party: Sponsor-Investigator, Dr. Tarit Saha, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ANAE-233-13
Record Dates: First submitted 2015-12-03; First posted 2016-03-03 (Estimated); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- slow sternal retraction (Experimental): sternal retraction (which is required for exposure of the heart during coronary artery bypass graft surgery) will be performed gradually over 15 minutes
  Interventions: Procedure: slow sternal retraction
- standard sternal retraction (No Intervention): sternal retraction will be performed as per standard practice (sternum opened rapidly over 30 sec.)

INTERVENTIONS:
Procedure: slow sternal retraction — the sternal retraction (which always need to be performed for coronary artery bypass graft surgery) will be achieved over 15 min instead of the usual 30 sec
  Other Names: slow retraction
  Arms: slow sternal retraction

SUMMARY:
In North America, almost ½ million people undergo coronary artery bypass graft surgery annually and over 1/3rd develop chronic chest pain. The current study will randomize cardiac surgery patients to undergo slow sternal retraction for heart exposure (over 15 min.) versus standard-of-care (sternal opening over 30 seconds) and examine the incidence and severity of chronic post-sternotomy pain (CPSP) and quality-of life 3, 6 and 12 months post-operatively. The severity of acute post-operative pain will also be measured. Increased retraction time reduces forces required, which should translate to reduced nerve/tissue damage. If effective, this simple change in practice could be readily implemented with a major impact for patients and the health care system overall.

DETAILED DESCRIPTION:
The overall objective of the current investigation is to determine whether increasing the time to sternal retraction to 15 minutes (from the standard ~30 sec), will result in reduced acute and chronic post-sternotomy pain and an improved quality of life. The hypothesis here is that increased time to sternal retraction will result in: reduced required force, less physical trauma, less inflammation, and less nerve damage. Specifically, the hypothesis is that slow steady sternal retraction (occurring over 15 minutes) will 1) reduce the incidence of CPSP by 40% 2) reduce the severity of acute postoperative pain by at least 20-30% and 3) significantly improve quality of life 6 months postoperatively.

The current investigation will be a prospective blinded, randomized, controlled trial. Following institutional ethics approval and signed consent, eligible patients scheduled for elective coronary artery bypass graft surgery will be randomly assigned (stratified by gender and surgeon to ensure equality between groups) either to the Standard group (in which sternal retraction occurs over ~30s) or the Slow group in which sternal retraction occurs over 15 minutes. Patients and research personnel performing the postoperative assessments will remain blinded to group assignment until conclusion of the investigation. All other intra-operative variables will be performed as per standard practice by the cardiac surgeons at Kingston General Hospital. The extent of sternal retraction will be to the surgeon's discretion to enable appropriate exposure of the heart to allow safe conduct of the operation but it will be recorded in all cases.

The primary outcome measure will be the incidence of chronic post-sternotomy chest pain 6 months following CABG with median sternotomy. However, we will also measure the incidence of CPSP at 3 and 12 months to determine the trajectory. Secondary outcomes will include: Pain intensity (numeric rating scale-NRS) of chest pain (which differs from preoperative) at rest and while coughing daily while in hospital until discharge and at 1 week postoperatively. Analgesic consumption (morphine equivalents) daily while in hospital until discharge, 1 week post-operatively and then at 3, 6, and 12 months postoperatively. Intra-operative data will include time from initiation to full retraction, latency from full retraction to sternal closure, width of sternal opening at full retraction. Pain quality, quality of life, and pain interference with daily function at 3, 6 and 12 months post-operatively. All assessments following discharge from the hospital will be via telephone calls from a research nurse blinded to randomization assignment. In-hospital assessments will also be done by a research nurse blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary artery bypass graft surgery
* understand written informed consent
* ASA I,II or III

Exclusion Criteria:

* revision cardiac surgery
* current alcohol/substance abuse
* pre-existing chronic pain requiring chronic analgesic use
* rest pain in proposed surgical area preoperatively
* chronic steroid use
* inability to perform postoperative assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic post-sternotomy pain | 6 months postoperatively
  incidence of chronic post-sternotomy pain 6 months following coronary artery bypass graft surgery

SECONDARY OUTCOMES:
Incidence of chronic post-sternotomy pain | 3 and 12 months postoperatively
  incidence of chronic pain
severity of chronic postoperative pain | 3 months. 6 months, 1 year
  pain on NRS scale
severity of acute postoperative pain at rest and with coughing | daily while an inpatient up to 1 week postoperatively
  pain on NRS scale
analgesic consumption | daily while an inpatient up to 1 week postoperatively, 1 week postoperatively, 3, 6 and 12 months postoperatively
quality of life with the Modified Brief Pain Inventory (BPI) | 3, 6, 12 months postoperatively
pain quality with the Douleur Neuropathique Questionnaire (DN4) | 3, 6 and 12 months postoperatively
pain quality with the McGill Pain Questionnaire-short form (MPQ-SF) | 3, 6 and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Tarit Saha, MD, FRCPC, Principal Investigator — Queen's University/Kingston General Hospital; Dimitri Petsikas, MD, FRCSC, Principal Investigator — Queen's University/ Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No